CLINICAL TRIAL: NCT01804829
Title: A Multi-Center, Randomized, Prospective, Open-Label Phase III Study to Evaluate the Efficacy, Safety and Pharmacokinetics of Hepatitis C Immune Globulin Intravenous (Human), Civacir®, in Orthotopic Liver Transplant Recipients
Brief Title: Civacir® Polyclonal Immune Globulin (IgG) to Prevent Hepatitis C Virus (HCV) Recurrence in Liver Transplant Patients.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biotest Pharmaceuticals Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 988
Record Dates: First submitted 2013-03-04; First posted 2013-03-05 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis C Infection; Viruses; Hepatocellular Carcinoma; Hepatitis, Viral, Human; Liver Cirrhosis
Keywords: HCV Liver Transplant Immunoglobulin PCR SVR
MeSH Terms: conditions — Hepatitis C; Virus Diseases; Carcinoma, Hepatocellular; Hepatitis, Viral, Human; Liver Cirrhosis | interventions — hepatitis C immune globulin, human; Immunoglobulin G

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Observational Control (No Intervention): Subjects who attain HCV RNA <100 IU/ml and are randomized to the control arm will receive standard post-transplant immunosuppressant therapy and be followed for a 34 week period.
- Civacir® 10% at 200 mg/kg dose (Experimental): Subjects who attain HCV RNA <100 IU/ml and are randomized to the Civacir 200 mg/kg treatment arm will receive Civacir® before liver transplant, followed by 15 infusions over a 10 week regimen, with standard post-transplant immunosuppressant therapy. Civacir® treated subjects will be followed up to 34 weeks post-transplant.
  Interventions: Biological: Civacir® 10%
- Civacir® 10% at 300 mg/kg dose (Experimental): Subjects who attain HCV RNA <100 IU/ml and are randomized to the Civacir® 300 mg/kg treatment arm will receive Civacir® before liver transplant, followed by 15 infusions over a 10 week regimen, with standard post-transplant immunosuppressant therapy. Civacir® treated subjects will be followed up to 34 weeks post-transplant.
  Interventions: Biological: Civacir® 10%

INTERVENTIONS:
Biological: Civacir® 10% — The active ingredient is Human Immunoglobulin G (IgG) which is a normal constituent purified from human source plasma containing a diversity of antibodies targeting the Hepatitis C Virus.
  Other Names: Civacir®; Hepatitis C Immune Globulin Intravenous (Human); human polyclonal immune globulin (IgG); HCIg
  Arms: Civacir® 10% at 200 mg/kg dose; Civacir® 10% at 300 mg/kg dose

SUMMARY:
The purpose of this study is to test the safety and efficacy of Civacir® to prevent the recurrence of Hepatitis C Virus (HCV) after liver transplant.

DETAILED DESCRIPTION:
Civacir® 10%, Hepatitis C Immune Globulin Intravenous (Human) is a high-titer human polyclonal immune globulin (IgG) containing a diversity of antibodies that target and bind the hepatitis C virus (HCV) to prevent infection. Subjects who reduce their viral load to less than 100 IU/ml HCV RNA through up to 24 weeks of antiviral therapy prior to liver transplant are enrolled in the study. There is no requirement to reach undetectable virus prior to transplant as the function of Civacir® is to neutralize any remaining virus in circulation.

Subjects randomized to Civacir® treatment arms receive study drug infusions starting on the day of liver transplant followed by 15 doses over a 10 week period to prevent the recurrence of quantifiable Hepatitis C Virus (HCV) after liver transplant. The study will evaluate dosing arms ranging from 200 mg/kg to 300 mg/kg compared to a control arm. For the primary endpoint, efficacy is defined as persistent viral load suppression maintaining HCV RNA levels below the lower limit of quantitation as determined by central laboratory Polymerase Chain Reaction (PCR) at 22 weeks post-liver transplant and then at 34 weeks post-liver transplant to demonstrate durability of effect.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained prior to any study-specific assessments and within 3 months (reconsent) of orthotopic liver transplantation (OLT).
* HCV Genotype 1 through 6 Infection.
* Subjects in the beginning of a new antiviral therapy regimen (regardless of prior treatment failures) for up to and including 24 weeks prior to the day of OLT.
* Most recent evidence within the last 4 weeks that HCV RNA is <100 IU/mL. Subjects may be randomized based on local lab HCV RNA.
* Male and female subjects (age 18-80 years).
* Subject weight under 250 pounds.
* Stable patient in a condition which in the opinion of the investigator would permit safe participation in the study.

Exclusion Criteria:

* Re-transplantation due to viral recurrence.
* Positive HIV or HBV test within 90 days prior to transplantation.
* Most recent PCR test indicating HCV RNA ≥100 IU/mL within 4 weeks of OLT.
* Subjects having received organs from HCV positive donors.
* Serum creatinine level >2.5 times the upper limit of normal or advanced renal disease at screening.
* Pregnancy or single contraceptive measure or lactation period (females only).
* Known intolerance to immunoglobulins or comparable substances (e.g. vaccination reaction).
* Known absolute Immunoglobulin A (IgA) deficiency.
* Known intolerance to proteins of human origin.
* Participation in another clinical trial within 90 days before signing Informed Consent Form (ICF) or during the study (observational/ non-interventional and 988 studies allowed), and/or previous participation in 988 study (except for Study 988 screen failures).
* Active drug and/or alcohol abuse.
* Inability or lacking motivation to participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-06; Primary Completion 2016-02 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Determine the efficacy of Civacir® in preventing post-transplant HCV recurrence at 22 weeks post transplant | 22 weeks
  The primary objective is to assess the effect of administering Civacir® anti-HCV immunoglobulin therapy on prevention of orthotopic liver transplant (OLT) HCV recurrence, as measured by the proportion of subjects with unquantifiable HCV RNA levels at 22 weeks post-OLT, compared to the control group (not treated with Civacir® and considered standard of care).

SECONDARY OUTCOMES:
Determine the efficacy of Civacir® in preventing post-transplant HCV recurrence at 4 and 34 weeks post transplant | 34 weeks
  Evaluate the proportion of subjects with unquantifiable HCV RNA, as measured quantitatively by PCR at 4 and 34 weeks post-OLT, for assessing the durability of effect.

OTHER OUTCOMES:
Determine the biochemical response of Civacir® in preventing post-transplant HCV recurrence at 22 and 34 weeks post transplant | 34 weeks
  Evaluate the biochemical response at 22 and 34 weeks post-transplant: the proportions of subjects with normal ALT, AST, total bilirubin and alkaline phosphates at 22 and 34 weeks.
Evaluate the safety of Civacir® in preventing post-transplant HCV recurrence up to 34 weeks post transplant | 34 weeks
  Evaluate the safety of Civacir® in the treatment of subjects with HCV undergoing liver transplantation by the number of adverse events including safety laboratory parameters.
Evaluate the pharmacokinetics of Civacir® up to 34 weeks post transplant | 34 weeks
  Evaluate the pharmacokinetics of Civacir® following intravenous infusion(s).

CONTACTS AND LOCATIONS:
Overall Officials: Norah Terrault, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (23):
- United States (23):
  - University of Southern California / Keck Hospital, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - University of Miami Miller School of Medicine, Miami, Florida
  - Florida Hospital Transplant Institute, Orlando, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University School of Medicine, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Ochsner Medical Center, New Orleans, Louisiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lahey Hospital, Burlington, Massachusetts
  - NYU Langone Medical Center, New York, New York
  - The Mount Sinai Medical Center, New York, New York
  - Columbia University College of Physicians and Surgeons, New York, New York
  - Oregon Health & Science University, Portland, Oregon
  - Methodist University Hospital, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - Advanced Liver Therapies / St. Luke's Episcopal Hospital, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Houston Methodist, Houston, Texas
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - University of Virginia Health System, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Everson GT, Terrault NA, Lok AS, Rodrigo del R, Brown RS Jr, Saab S, Shiffman ML, Al-Osaimi AM, Kulik LM, Gillespie BW, Everhart JE; Adult-to-Adult Living Donor Liver Transplantation Cohort Study. A randomized controlled trial of pretransplant antiviral therapy to prevent recurrence of hepatitis C after liver transplantation. Hepatology. 2013 May;57(5):1752-62. doi: 10.1002/hep.25976. Epub 2013 Jan 17. PMID 22821361
- [Background] Davis GL, Nelson DR, Terrault N, Pruett TL, Schiano TD, Fletcher CV, Sapan CV, Riser LN, Li Y, Whitley RJ, Gnann JW Jr; Collaborative Antiviral Study Group. A randomized, open-label study to evaluate the safety and pharmacokinetics of human hepatitis C immune globulin (Civacir) in liver transplant recipients. Liver Transpl. 2005 Aug;11(8):941-9. doi: 10.1002/lt.20405. PMID 16035063